CLINICAL TRIAL: NCT01587833
Title: WEUKBRE5559: IMI PROTECT (Work Package 2): Use of Benzodiazepines and Risk of Hip/Femur Fracture
Brief Title: WEUKBRE5559: IMI PROTECT: Benzodiazepines & Fracture
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116440
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Anxiety Disorders
Keywords: Benzodiazepines; hip/femur fracture
MeSH Terms: conditions — Anxiety Disorders | interventions — Benzodiazepines

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with a diagnosis of hip or femur fracture: All patients of the study population with a record/diagnosis of a first fracture of the hip or femur during the study period regardless of whether they have a history of past fractures. When the patient has a history of hip or hip/femur fracture, a minimum of 12 months should have elapsed between the two episodes for a current fracture to be considered a new event.
  Interventions: Drug: Benzodiazepine (BZD) use, defined by ATC codes
- Patients without a diagnosis of hip or femur fracture: All patients of the study population without a record/diagnosis of a fracture of the hip or femur during the study period
  Interventions: Drug: Benzodiazepine (BZD) use, defined by ATC codes

INTERVENTIONS:
Drug: Benzodiazepine (BZD) use, defined by ATC codes — BZD prescription during the study period between January 1, 2001 and December 31, 2009

SUMMARY:
The studies described in this protocol are all performed within the framework of PROTECT (Pharmacoepidemiological Research on Outcomes of Therapeutics by a European ConsorTium) Workpackage 2 and Workgroup 1. Primary aim of these studies is to develop, test and disseminate methodological standards for the design, conduct and analysis of Pharmacoepidemiological (PE) studies applicable to different safety issues and using different data sources. To achieve this, results from PE studies on five key adverse events (AEs) performed in different databases will be evaluated. Therefore, emphasis will be on the methodological aspects of the studies in this protocol and not on the clinical consequences of the association under investigation.

Benzodiazepines (BZDs) are one of the therapeutic groups most widely used, mainly indicated as hypnotics and anxiolytics. Guidelines recommend treatment courses not exceeding 4-6 weeks. However, long-term treatment is highly prevalent, particularly in older people with a prevalence ranging from 15 to 30%. However, treatment is often taken as needed.

Hip/femur fractures are a major cause of morbidity and mortality, impair quality of life and impose a considerable economic burden. Among people aged 50 years and older, a case-fatality rate of 20% is associated within the first year.

The relationship between benzodiazepines and hip fractures remains controversial. Psychotropic medication has been traditionally associated with hip fractures. Among psychotropic medication, long elimination half-life benzodiazepines were found to increase the risk of hip fractures in a case-control study published in the late eighties. Since then, several investigations have been performed, mostly in older patients focusing on the relationship between benzodiazepines and hip fractures, and between benzodiazepines and falls as a mechanism underlying this effect. A review performed in 2003, which included 11 epidemiological studies, reported that results were not always consistent. Seven out of eight cohort and population based case-control studies, found an association, but different results were reported according to benzodiazepines' half-life. In four hospital-based case-control studies no association between benzodiazepines use and hip fracture has been described. Data on dosing was only included in three of the studies, and once more results were not conclusive. Results ranged from no effect to an increased risk with high dose regimens. Results from subsequent succeeding studies have also shown contradictions, with no association reported in one of the studies, and an association described for the short-term use of short half-life, high-potency benzodiazepines.

Even though there is epidemiological evidence suggesting that the use of benzodiazepines increases the risk of hip fractures, problems rise with the definition of benzodiazepine exposure, or biases such as confounding by indication and the control for confounders. These remain unresolved topics that should be addressed in future studies. In the present protocol, it is proposed to further asses the risk of hip/femur fractures associated with benzodiazepines using different study designs in different primary databases, and to compare the results in order to evaluate the impact of design and population differences on the outcome of the study association.

The objective of this study is to assess the association between benzodiazepines use and hip/femur fracture with different study designs (descriptive, cohort, nested case-control, case crossover and self control case series) across different primary care databases (Bavarian, Mondriaan, National Databases (Denmark), General Practice Research Database (GPRD), Base de Datos para la Investigación Farmacoepidemiologica en Atencion Primaria (BIFAP) and The Health Improvement Network (THIN)) and to compare the results between databases, across designs to evaluate the impact of design/database/population differences on the outcome of the studied association.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have at least one year of enrolment with the GP
* All patients who are at least 18 years of age
* All patients who have at least one benzodiazepine prescription

Exclusion Criteria:

* Patients with a benzodiazepine prescription within 6 months prior to study start
* Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all patients included in the period of valid data collection from the following data bases: Bavarian, Mondriaan, National Databases (Denmark), GPRD, BIFAP and THIN. The study period will be defined from January 1, 2001 to December 31, 2009.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incident hip/femur fracture defined by ICPE-2 codes in BIFAP/Mondriaan, Read codes in GPRD/THIN and ICD-10 codes in Bavarian database | Up to nine years following drug exposure

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline